CLINICAL TRIAL: NCT04393844
Title: Comparison of Success Rate of Catheter Insertion by the Presence of Obturator During Peripherally Inserted Central Venous Catheter in Pediatric Patient Undergoing General Anesthesia; Prospective Randomized Controlled Study
Brief Title: The Success Rate of Catheter Insertion by the Presence of Obturator During Peripherally Inserted Central Venous Catheter
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Hee-Soo Kim, Professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 2004-206-1120
Record Dates: First submitted 2020-05-14; First posted 2020-05-19 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Central Venous Catheters

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- with obturator (Placebo Comparator): A group using an obturator when performing peripherally inserted central venous catheterization in children under 18 years of age under general anesthesia.
  Interventions: Other: turbo-ject PICC set
- without obturator (Experimental): A group that does not use an obturator when performing peripherally inserted central venous catheterization in children under 18 years of age under general anesthesia.
  Interventions: Other: turbo-ject PICC set

INTERVENTIONS:
Other: turbo-ject PICC set — The turbo-ject PICC set, which will be used in this study, is the set for peripherally inserted central catheterization. In this study, we will see the difference according to the presence or absence of the hydrophilic coated stiffening obturator included in this turbo-ject PICC set.

SUMMARY:
In pediatric patients under the age of 18 who undergo surgery under general anesthesia, when inserting peripherally inserted central venous catheterization, the group that inserts the catheter with the obturator and the group that inserts the catheter without the obturator is inserted into the appropriate position.

DETAILED DESCRIPTION:
In pediatric patients under the age of 18 who undergo surgery under general anesthesia, when inserting peripherally inserted central venous catheterization, the group that inserts the catheter with the obturator and the group that inserts the catheter without the obturator is inserted into the appropriate position.

There is no study confirming the probability of being placed in the central vein at a time when the catheter is inserted without the obturator, and there is no study comparing the clinical effect by dividing the case with the obturator and the obturator. In children, the blood vessels are small and there is a high probability that they cannot be located in the central vein when the peripheral vein is inserted.

Therefore, when a peripheral implanted central venous tube is inserted into a pediatric patient under general anesthesia under 18 years of age, the probability that the catheter is inserted without using an obturator will be located in the central vein at a time rather than using an obturator to insert the catheter. It could help pediatric patients to manage anesthesia and post-surgical care by reducing potential complications from using obturator.

ELIGIBILITY:
Inclusion Criteria:

* Children under 18 years of age undergoing general anesthesia surgery at Seoul National University Hospital
* ASA class I, II
* If the legal guardian voluntarily consents after the explanation of the research

Exclusion Criteria:

* Patients with a history of heart surgery or a history of congenital heart disease
* Patients with hemodynamically unstable or massive bleeding and shock
* Infection or systemic infection is suspected
* Patients who have a blood clotting disorder
* Abnormal cases when the vessel to be inserted is confirmed by ultrasound
* the cases that the researcher determines that it is inappropriate

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 65 (Actual)
Dates: Start 2020-06-02 (Actual); Primary Completion 2022-04-17 (Actual); Study Completion 2023-07-15 (Estimated)

PRIMARY OUTCOMES:
Success rate at one time | confirmation through ultrasound procedure completed
  Success rate to place into the central vein without additional treatment at one time

SECONDARY OUTCOMES:
Number of insertion attempts | during procedure
  Number of insertion attempts to place into the central vein
Number of additional manipulation | during procedure
  Number of additional manipulation to place into the central vein
type of additional manipulation | during procedure
  type of additional manipulation to place into the central vein
the location of catheter in case of the malposition at one time | confirmation through ultrasound procedure completed
  the location of catheter in case of the malposition at one time
final success rate | procedure
  final success rate based on confirming in postoperative chest x-ray
final catheter location | procedure
  final catheter location confirming in postoperative chest X-ray
other complication | procedure
  other complication such as hematoma, vessel rupture, nonfunction, kinking of catheter

CONTACTS AND LOCATIONS:
Overall Officials: Hee-Soo Kim, MD, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Seoul, South Korea, South Korea

IPD SHARING:
Plan to Share IPD: No